CLINICAL TRIAL: NCT00516477
Title: A Phase 1 Safety Study in Subjects With Leber Congenital Amaurosis (LCA) Using Adeno-Associated Viral Vector to Deliver the Gene for Human RPE65 Into the Retinal Pigment Epithelium (RPE) [AAV2-hRPE65v2-101]
Brief Title: Safety Study in Subjects With Leber Congenital Amaurosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAV2-hRPE65v2-101; 2006-6-4787 (Other: Children's Hospital of Philadelphia IRB)
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Leber Congenital Amaurosis
Keywords: Adeno-Associated Virus (AAV); Leber Congenital Amaurosis; Gene transfer
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- dose cohort 1 (Experimental): 1.5E10 vector genomes voretigene neparvovec-rzyl in 150 microliters administered subretinally
  Interventions: Biological: voretigene neparvovec-rzyl
- dose cohort 2 (Experimental): 4.8E10 vector genomes voretigene neparvovec-rzyl in 150 microliters administered subretinally
  Interventions: Biological: voretigene neparvovec-rzyl
- dose cohort 3 (Experimental): 1.5E11 vector genomes voretigene neparvovec-rzyl in 300 microliters administered subretinally
  Interventions: Biological: voretigene neparvovec-rzyl

INTERVENTIONS:
Biological: voretigene neparvovec-rzyl — Subjects will be dosed unilaterally (one eye) beginning with the lowest dose. Subjects will be injected with AAV2-hRPE65v2 by means of a subretinal injection. Dose escalation to the next cohort will be dependent on assessment of the safety data by the DSMB out to at least 4 weeks following the injection. Because there is a delay between time of delivery of AAV2 and the peak transgene expression there will be a delay of six weeks between all subjects.
  Other Names: AAV2-hRPE65v2

SUMMARY:
The purpose of this study is to determine whether gene transfer will be safe and effective in the treatment of Leber Congenital Amaurosis (LCA).

DETAILED DESCRIPTION:
Leber Congenital Amaurosis (LCA)is a severe early onset retinal degeneration. Diagnosis is usually made during the first few months of life in infants who present with severely impaired vision, abnormal eye movements (nystagmus) and abnormal electroretinograms (ERG) indicating decreased retinal function. There is an inevitable progression to total blindness in these individuals due to death of photoreceptor cells. There is presently no treatment for this disease. The primary objective of this study is to determine the safety and tolerability of subretinal administration of AAV2-hRPE65v2 to subjects with LCA due to confirmed biallelic RPE65 mutations. The secondary objective is to assess the objective clinical measures of efficacy in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of any ethnic group are eligible for participation in this study, providing they meet the following criteria:

  1. Must be willing to adhere to protocol and companion protocol for long-term follow-up as evidenced by written informed consent or parental permission and subject assent.
  2. Adults and children diagnosed with LCA.
  3. Molecular diagnosis of LCA due to RPE65 mutations (homozygotes or compound heterozygotes) by a CLIA-approved laboratory.
  4. Age eight years old or older at the time of administration.
  5. Visual acuity ≤ 20/160 or visual field less than 20 degrees in the eye to be injected.

Exclusion Criteria:

SUBJECTS WILL NOT BE EXCLUDED BASED ON THEIR GENDER, RACE OR ETHNICITY.

Subjects who meet any of the following conditions are excluded from the clinical study:

1. Unable or unwilling to meet requirements of the study.
2. Participation in a clinical study with an investigational drug in the past six months.
3. Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints (for example, glaucoma, corneal or lenticular opacities).
4. Lack of sufficient viable retinal cells as determined by non-invasive means, such as optical coherence tomography (OCT) and/or ophthalmoscopy. Specifically, if indirect ophthalmoscopy reveals less than 1 disc area of retina which is not involved by complete retinal degeneration (indicated by geographic atrophy, thinning with tapetal sheen, or confluent intraretinal pigment migration), these eyes will be excluded. In addition, in eyes where optical coherence tomography (OCT) scans of sufficient quality can be obtained, areas of retina with thickness measurements less than 100 um, or absence of neural retina, will not be targeted for delivery of AAV2-hRPE65v2.
5. Complicating systemic diseases or clinically significant abnormal baseline laboratory values. Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter ocular function. Examples are malignancies whose treatment could affect central nervous system function (for example, radiation treatment of the orbit; leukemia with CNS/optic nerve involvement). Also excluded would be subjects with immuno-compromising diseases, as there could be susceptibility to opportunistic infection (such as CMV retinitis). Subjects with diabetes or sickle cell disease would be excluded if they had any manifestation of advanced retinopathy (e.g. macular edema or proliferative changes). Subjects with juvenile rheumatoid arthritis could be excluded due to increased infection risk after surgery due to poor wound healing. Subjects who are positive for hepatitis B, C, and HIV will be excluded.
6. Prior ocular surgery within six months.
7. Known sensitivity to medications planned for use in the peri-operative period.
8. Individuals of childbearing potential who are pregnant or unwilling to use effective contraception for the duration of the study.
9. Any other condition that would not allow the potential subject to complete follow-up examinations during the course of the study and, in the opinion of the investigator, makes the potential subject unsuitable for the study.
10. Subjects will be excluded if immunological studies show presence of neutralizing antibodies to AAV2 above 1:1000.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-09 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests. | Visual function will be measured at designated intervals from baseline visits through 5 years as stated in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Spark Therapeutics, Inc.
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Acland GM, Aguirre GD, Ray J, Zhang Q, Aleman TS, Cideciyan AV, Pearce-Kelling SE, Anand V, Zeng Y, Maguire AM, Jacobson SG, Hauswirth WW, Bennett J. Gene therapy restores vision in a canine model of childhood blindness. Nat Genet. 2001 May;28(1):92-5. doi: 10.1038/ng0501-92. PMID 11326284
- [Background] Acland GM, Aguirre GD, Bennett J, Aleman TS, Cideciyan AV, Bennicelli J, Dejneka NS, Pearce-Kelling SE, Maguire AM, Palczewski K, Hauswirth WW, Jacobson SG. Long-term restoration of rod and cone vision by single dose rAAV-mediated gene transfer to the retina in a canine model of childhood blindness. Mol Ther. 2005 Dec;12(6):1072-82. doi: 10.1016/j.ymthe.2005.08.008. Epub 2005 Oct 14. PMID 16226919
- [Background] Bennett J, Maguire AM, Cideciyan AV, Schnell M, Glover E, Anand V, Aleman TS, Chirmule N, Gupta AR, Huang Y, Gao GP, Nyberg WC, Tazelaar J, Hughes J, Wilson JM, Jacobson SG. Stable transgene expression in rod photoreceptors after recombinant adeno-associated virus-mediated gene transfer to monkey retina. Proc Natl Acad Sci U S A. 1999 Aug 17;96(17):9920-5. doi: 10.1073/pnas.96.17.9920. PMID 10449795
- [Result] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Result] Maguire AM, High KA, Auricchio A, Wright JF, Pierce EA, Testa F, Mingozzi F, Bennicelli JL, Ying GS, Rossi S, Fulton A, Marshall KA, Banfi S, Chung DC, Morgan JI, Hauck B, Zelenaia O, Zhu X, Raffini L, Coppieters F, De Baere E, Shindler KS, Volpe NJ, Surace EM, Acerra C, Lyubarsky A, Redmond TM, Stone E, Sun J, McDonnell JW, Leroy BP, Simonelli F, Bennett J. Age-dependent effects of RPE65 gene therapy for Leber's congenital amaurosis: a phase 1 dose-escalation trial. Lancet. 2009 Nov 7;374(9701):1597-605. doi: 10.1016/S0140-6736(09)61836-5. Epub 2009 Oct 23. PMID 19854499
- [Result] Simonelli F, Maguire AM, Testa F, Pierce EA, Mingozzi F, Bennicelli JL, Rossi S, Marshall K, Banfi S, Surace EM, Sun J, Redmond TM, Zhu X, Shindler KS, Ying GS, Ziviello C, Acerra C, Wright JF, McDonnell JW, High KA, Bennett J, Auricchio A. Gene therapy for Leber's congenital amaurosis is safe and effective through 1.5 years after vector administration. Mol Ther. 2010 Mar;18(3):643-50. doi: 10.1038/mt.2009.277. Epub 2009 Dec 1. PMID 19953081
- [Result] Ashtari M, Cyckowski LL, Monroe JF, Marshall KA, Chung DC, Auricchio A, Simonelli F, Leroy BP, Maguire AM, Shindler KS, Bennett J. The human visual cortex responds to gene therapy-mediated recovery of retinal function. J Clin Invest. 2011 Jun;121(6):2160-8. doi: 10.1172/JCI57377. Epub 2011 May 23. PMID 21606598
- [Derived] Fischer MD, Simonelli F, Sahni J, Holz FG, Maier R, Fasser C, Suhner A, Stiehl DP, Chen B, Audo I, Leroy BP; PERCEIVE Study Group. Real-World Safety and Effectiveness of Voretigene Neparvovec: Results up to 2 Years from the Prospective, Registry-Based PERCEIVE Study. Biomolecules. 2024 Jan 17;14(1):122. doi: 10.3390/biom14010122. PMID 38254722
- [Derived] Melillo P, Pecchia L, Testa F, Rossi S, Bennett J, Simonelli F. Pupillometric analysis for assessment of gene therapy in Leber Congenital Amaurosis patients. Biomed Eng Online. 2012 Jul 19;11:40. doi: 10.1186/1475-925X-11-40. PMID 22812667